CLINICAL TRIAL: NCT05531851
Title: Effects of Instrument Assisted Soft Tissue Mobilization on Delayed Onset Muscle Soreness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Harran University (Other)
Responsible Party: Principal Investigator, İSMAİL PALALI, Lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SaglikBilimleriU-63
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Musculoskeletal Pain; Soreness, Muscle; Musculoskeletal Disorder
Keywords: Delayed onset muscle soreness, Instrument-assisted soft tissue mobilization, recovery, eccentric exercise
MeSH Terms: conditions — Musculoskeletal Pain; Myalgia; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group. (Experimental): İnstrument-assisted soft tissue mobilization will be applied after the delayed onset muscle soreness induction protocol
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization
- Control Group (No Intervention): Delayed onset muscle soreness generation protocol will be applied

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — For IASTM treatment, IASTM soft tissue mobilization blade to apply the treatment used. It is a stainless steel shaped metal tool with beveled edges. The researcher, with a 30° angled tool, at a speed of 120 BPM, in the direction of the fibers of the m.biceps brachii muscle.
  He applied it with a light pressure by intervening with his weight. Researcher during treatment used a metronome to ensure consistent speed and adjusted the instrument angle before each subject's treatment.
  calibrated with a protractor. The application took 8 minutes and the instrument was comfortable on the skin.
  Arms: Experiment group.

SUMMARY:
The aim of our study is to investigate the effect of instrument assisted soft tissue mobilization therapy on delayed onset muscle soreness

DETAILED DESCRIPTION:
Joint range of motion, pressure pain threshold, edema, isometric muscle strength measurement, visual pain scale, two-point discrimination, biochemical measurements (muscle damage in blood (serum creatine kinase (CC), lactate dehydrogenase (LDH), myoglobin, its effects on aspartate aminotransferase (AST) and alanine aminotransferase (ALT) and biomarkers of inflammation (interleukin-1 beta), Carbonic anhydrase III, and C-reactive protein, and at what time interval and after which treatment session in the process after delayed muscle pain formation. It is aimed to determine how it affects the parameters.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be between the ages of 18-35,
2. No fear of needles,
3. Having read and understood the Informed Voluntary Consent Form and agreeing to participate in the study.

Exclusion Criteria:

1. Having neurological or perception problems,
2. Having any cardiovascular, pulmonary and metabolic disease,
3. Any musculoskeletal injury in the last 6 months,
4. Having a history of pain and surgery in the upper extremity,
5. Participating in upper extremity weight training in the last 6 months,
6. Exercise, caffeine and alcohol consumption, and drug use up to 12 hours before the study were determined as

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Four days
  0-100 mm Visual Analogue Scale (VAS) to assess perceived muscle pain and muscle fatigue used. Visual Analog Scale on a straight line with a value of '0' means 'no pain/fatigue', A value of '100' is a scale that indicates 'severe pain/fatigue'. The pain felt by the participants and will be asked to mark the fatigue with an x on this line, Perceived pain both during rest and evaluated during active flexion-extension movement. Perceived fatigue is just rest.
  evaluated while in position.
Pressure-pain threshold measurement | Four days
  ll measurements were evaluated using an algometer while the participants were lying in the supine position.
  The forearm is at 90º pronation at the side of the body and the elbow is at 0º extension.
  point application. reference point for measurement; three centimeters below the medial epicondyle While determining the pressure point, it was chosen as six centimeters above this reference point. measuring Before starting, a control trial was made, and the participant was asked to say "yes" as soon as they felt "discomfort" or "pain".
  required is specified.fatigue used. Visual Analog Scale on a straight line with a value of '0' means 'no pain/fatigue', A value of '100' is a scale that indicates 'severe pain/fatigue'. The pain felt by the participants and will be asked to mark the fatigue with an x on this line, Perceived pain both during rest and evaluated during active flexion-extension movement. Perceived fatigue is just rest.
  evaluated while in position.
Circumference measurement | Four days
  Edema in the biceps brachii muscle will be evaluated by measuring the circumference Non-flexible tape measure for measurement used. The measurement was taken 3 cm above (lower arm) and 12 cm above (upper arm) elbow crease.
  Two measurements were made from both points and recorded by taking the average. Participant standing, relaxed The measurement was made in the position and the arm was near the body. The marked point is at the bottom line of the tape measure.
  measurement was carried out.
Joint range of motion measurement | Four days
  Joint range of motion measurement will be made with a digital goniometer. loosely rested. Participants try to touch their shoulders with their palms for the EHAFLEX measurement.
  fully flexed the elbows, and fully extended the elbow joint for the EHAEXT measurement.
  tried to bring Measurements were recorded by repeating 2 times and taking the average.Non-flexible tape measure for measurement used. The measurement was taken 3 cm above (lower arm) and 12 cm above (upper arm) elbow crease.
  Two measurements were made from both points and recorded by taking the average. P
Isometric muscle strength | Four days
  Isometric muscle strength of elbow flexor muscles was evaluated by hand dynamometer. Participant elbow Seated in chair with forearm supinated at 90 degrees of flexion. Flexor of the forearm by placing it on the face proximal to the styloid process and flexing the elbow of the participant for 5 seconds.
  direction was requested. (maximum voluntary isometric contraction) and movement A force was applied in the opposite direction by the evaluator. 3 measurements were made at 30 second intervals and recorded by taking the average.
Two-point discrimination | Four days
  In our study, this measurement was made with a disc-criminator. This tool is embedded at varying intervals each It consists of two plastic discs containing rods. The distance between the bars varies from 1mm to 25mm.
  The value that the subjects felt as two points was recorded.
Liver enzymes (aminotransferases) | Four days
  The general name of these enzymes, which are specific to the liver and are frequently used to determine liver damage, are aminotransferases and consist of ALT, AST, Alkaline Phosphatase, Gamma Glutamyl Transpeptidase. ALT and especially AST are synthesized in skeletal and cardiac muscle, Gamma Glutamyl Transpeptidase in kidneys, Alkaline Phosphatase in bones and intestinal epithelial cells. Increases in ALT and AST levels are proportional to the level of cell damage in the body, and therefore, they are biochemical markers that are important in the progression of the damage or in the follow-up of the healing process. In heavy exercises, increases in AST and ALT enzyme levels are observed depending on the duration and intensity of the exercise.
Creatine kinase | Four days
  Serum CC is the intramuscular enzyme responsible for keeping ATP at the appropriate level during muscle contraction. In addition, it is the most valid protein that increases after exercise as the most important marker of muscle damage. An increase in the serum CC level indicates that the membrane surrounding the muscle cell is ruptured or its permeability is increased. The peak time of serum CC, which increases after exercise, varies depending on the type, intensity and duration of exercise. In general, it was stated that serum CC level started to rise after exercise, reached its highest level after 24 hours and continued for 48 hours.
Lactate dehydrogenase | Four days
  Another enzyme used to assess muscle damage is lactate dehydrogenase (LDH), which catalyzes the conversion of pyruvate to lactate in anaerobic glycolysis. In muscle damage after exercise, serum LDH level reaches its highest value in the first 6 hours and returns to its pre-exercise basal level 24-72 hours later.
Myoglobin | Four days
  It is a low-molecule protein found in heart and skeletal muscle and provides storage of oxygen and transport to mitochondria in the muscle cell. There are three different isoforms of myoglobin in skeletal muscle, and its secretion increases as a result of the deterioration of protein structures due to muscle damage after heavy exercises. After muscle damage, myoglobin level increases within 2 hours, reaches its highest value in 6-9 hours and returns to normal in 24-36 hours.
Interleukin-1 beta | Four days
  It is a low-molecule protein found in heart and skeletal muscle and provides storage of oxygen and transport to mitochondria in the muscle cell. There are three different isoforms of myoglobin in skeletal muscle, and its secretion increases as a result of the deterioration of protein structures due to muscle damage after heavy exercises. After muscle damage, myoglobin level increases within 2 hours, reaches its highest value in 6-9 hours and returns to normal in 24-36 hours.
C reactive protein | Four days
  CRP is another generally accepted marker of inflammation and is synthesized by the liver in response to high plasma levels of IL-6 in the body. CRP level is significantly increased in acute myocardial infarction, stress, trauma, infection, inflammation, post-surgery or neoplastic proliferation. The increase in CRP in muscle damage and inflammation that occurs after exercise begins within 6-8 hours and reaches its peak levels within 24-48 hours. However, studies give conflicting information about whether the CRP level will increase with exercise. These results suggest that more research is needed to fully understand the effects of plasma CRP response after vigorous exercise.
Carbonic anhydrase III | Four days
  Carbonic anhydrase III (CAIII) is a member of a multigene family (at least six separate genes are known) that encode carbonic anhydrase isozymes. These carbonic anhydrases are a class of metalloenzymes that catalyze the reversible hydration of carbon dioxide and are differentially expressed in a number of cell types.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Palalı, PhD (c), Principal Investigator — Harran University
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided